CLINICAL TRIAL: NCT00497978
Title: The Effect of Taurine on Morbidity and Mortality in the Elderly Hip Fracture Patient
Acronym: TAUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Responsible Party: Principal Investigator, Alexander P.J. Houdijk, MD, PhD, surgeon, Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TAUP03.04.07/2
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Insulin Resistance; Elderly Patient; Oxidative Stress
MeSH Terms: conditions — Insulin Resistance | interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): taurine will be given per capsule
  Interventions: Dietary Supplement: taurine
- 2 (Placebo Comparator): placebo capsules containing microcrystalline cellulose will be given
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: taurine — 6 grams of taurine will be given each day in capsules, starting the day of admission till the sixth postoperative day
  Arms: 1
Dietary Supplement: placebo — a similar amount of placebo will be given each day in capsules, starting the day of admission till the sixth postoperative day
  Arms: 2

SUMMARY:
The purpose of this study is to reduce the postoperative morbidity and mortality in the elderly hip fracture patient, by giving them taurine peri-operatively.

DETAILED DESCRIPTION:
Rationale: A growing medical concern is the increase in the number of very old patients, especially the patients undergoing hip fracture surgery are rapidly increasing in numbers. Hip surgery in these old patients induces serious morbidity and gives rise to excessive mortality rates. Studies with perioperative nutritional interventions performed within this population have shown improved clinical outcome, but were not well controlled and lack insight in the working mechanism. Therefore nutritional intervention studies are needed using a single nutrient. In trauma patients for instance it is known that the administration of glutamine (as a single amino acid) reduces morbidity, which is probably related to its antioxidant properties; reducing oxidative stress and insulin resistance. As an antioxidant the amino acid taurine has even greater potential providing benefit in several groups of patients. Elderly hip fracture patients have very low plasma levels of antioxidants which make them highly vulnerable for oxidative stress and related insulin resistance.In elderly patients with a hip fracture, it is hypothesized that taurine lowers oxidative stress and the related harmful insulin resistance, thereby reducing morbidity and mortality.

Objective: Our primary objective is to reduce morbidity and consequent mortality in the elderly hip fracture patient by the administration of taurine.

Study design: A double blind placebo controlled intervention study at the surgery department of the Medical Center Alkmaar. The study consists of three parts: 1. A dose finding study; 2. Main study: outcome study on morbidity and mortality; 3. A study on insulin resistance, parallel to the main study.

Study population: Patients of both genders and any ethnicity, who will undergo primary surgery for a hip fracture, aged over 75 years, will be eligible for the study.

Intervention: Patients will receive from the moment of admission oral administration of taurine (3g/day or 6g/day, depending on results of the dose finding study) or placebo.

Main study parameters/endpoints: The main study parameter is the morbidity and consequent mortality. The secondary study parameters are oxidative stress, postoperative insulin resistance, mitochondrial dysfunction in skeletal muscle and postoperative delirium.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The possible benefit of the study is related to the effect of taurine. Oral administration of taurine, as an antioxidant, perioperatively, can reduce morbidity and consequent mortality, reduce oxidative stress, counteract the postoperative insulin resistance and thereby enhance the clinical outcome of the elderly hip fracture patient. Research showed that taurine can be safely administered to humans and no adverse effects are reported. A part of the patients will undergo a hyperinsulinaemic euglycaemic clamp to assess hepatic and peripheral insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* age above 75 years old
* hip fracture with a primary indication for surgery
* having obtained his/her informed consent

Exclusion Criteria:

* participating in another clinical trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 236 (Actual)
Dates: Start 2008-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
morbidity and mortality | 1 year

SECONDARY OUTCOMES:
antioxidant/oxidant parameters and inflammatory mediators | 1 week
postoperative insulin resistance | 1 week
mitochondrial dysfunction in the skeletal muscle | 1 week
postoperative delirium incidence, duration and severity | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Alexander PJ Houdijk, MD, PhD, Principal Investigator — Medical Center Alkmaar
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Derived] Westhoff D, Witlox J, Koenderman L, Kalisvaart KJ, de Jonghe JF, van Stijn MF, Houdijk AP, Hoogland IC, Maclullich AM, van Westerloo DJ, van de Beek D, Eikelenboom P, van Gool WA. Preoperative cerebrospinal fluid cytokine levels and the risk of postoperative delirium in elderly hip fracture patients. J Neuroinflammation. 2013 Oct 7;10:122. doi: 10.1186/1742-2094-10-122. PMID 24093540
- [Derived] Witlox J, Slor CJ, Jansen RW, Kalisvaart KJ, van Stijn MF, Houdijk AP, Eikelenboom P, van Gool WA, de Jonghe JF. The neuropsychological sequelae of delirium in elderly patients with hip fracture three months after hospital discharge. Int Psychogeriatr. 2013 Sep;25(9):1521-31. doi: 10.1017/S1041610213000574. Epub 2013 May 7. PMID 23651760
- [Derived] Slor CJ, Witlox J, Jansen RW, Adamis D, Meagher DJ, Tieken E, Houdijk AP, van Gool WA, Eikelenboom P, de Jonghe JF. Affective functioning after delirium in elderly hip fracture patients. Int Psychogeriatr. 2013 Mar;25(3):445-55. doi: 10.1017/S1041610212001962. Epub 2012 Nov 30. PMID 23194775